CLINICAL TRIAL: NCT01435967
Title: Observational, Ecological, Database Study on Epidemiology of Hospitalisations With Rotavirus Gastroenteritis Confirmed in Children Aged ≤5 Years, and Any Impact in the Change From Lyophilised to Liquid Formulation of Rotarix™, in Belgium
Brief Title: Observational Study on Rotavirus Gastroenteritis Epidemiology, Impact of Lyophilised vs. Liquid Formulation of Rotarix™
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 114061
Record Dates: First submitted 2011-09-09; First posted 2011-09-19 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-03

CONDITIONS: Infections, Rotavirus
Keywords: Rotarix™; Observational; ecological
MeSH Terms: conditions — Rotavirus Infections | interventions — Data Collection

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Cohort A: Children aged <=5 years in Belgium, with opportunity to receive Rotarix, requiring hospitalisation during which rotavirus detection test was performed and with available results.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Data collected when only the lyophilised formulation of Rotarix was in use (which is considered as baseline) will be specifically compared to data collected post the introduction of the liquid formulation. The results will also be compared to available vaccine coverage data for those rotavirus vaccines being used in Belgium.

SUMMARY:
The aim of this study is to monitor any impact in the change from the lyophilised formulation to the liquid formulation of the Rotarix™ vaccine on hospitalisations for rotavirus gastroenteritis. This is planned to be assessed by comparing trends of hospitalisations due to laboratory confirmed rotavirus gastroenteritis in children <=5 years of age, before and after introduction of the liquid formulation of the vaccine in Belgium.

ELIGIBILITY:
Inclusion Criteria:

All subjects must satisfy ALL the following criteria at study entry:

* Child aged ≤5 years with opportunity to receive lyophilised or liquid formulation of Rotarix™;
* Hospitalised at one of the participating centres in Belgium;
* A stool sample has been provided for a rotavirus detection test during the study period;
* Laboratory test result of rotavirus is available.

Exclusion Criteria:

• None.

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children hospitalised due to laboratory confirmed rotavirus gastroenteritis in approximately 8 hospitals across Belgium.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2011-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Occurrence of rotavirus in hospitalised children aged ≤5 years during pre-introduction, introduction and post-introduction period of liquid formulation Rotarix™ | up to 2 years post-introduction of liquid formulation of Rotarix™.

SECONDARY OUTCOMES:
Occurrence of rotavirus detected by laboratory tests in children of various age, gender and location (centre and region). | up to 2 years post-introduction of liquid formulation of Rotarix™.
Occurrence of rotavirus detected by laboratory tests at a specific time (month and year). | up to 2 years post-introduction of liquid formulation of Rotarix™.
Occurrence of rotavirus detected by various types of rotavirus laboratory tests. | up to 2 years post-introduction of liquid formulation of Rotarix™.
Occurrence of rotavirus vaccination with a specific brand of vaccine (Rotarix and RotaTeq) among children ≤5 years of age in the Belgian population. | up to 2 years post-introduction of liquid formulation of Rotarix™.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- Belgium (8):
  - GSK Investigational Site, Antwerp
  - GSK Investigational Site, Bonheiden
  - GSK Investigational Site, Charleroi
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Hasselt
  - GSK Investigational Site, Ieper
  - GSK Investigational Site, Jette
  - GSK Investigational Site, Yvoir

REFERENCES:
- [Derived] Raes M, Strens D, Kleintjens J, Biundo E, Morel T, Vyse A. Epidemiological trends for hospital admissions for acute rotavirus gastroenteritis in Belgium following the introduction of routine rotavirus vaccination and the subsequent switch from lyophilized to liquid formulation of Rotarix. Epidemiol Infect. 2016 Oct;144(14):3017-3024. doi: 10.1017/S0950268816001151. Epub 2016 Jul 4. PMID 27373141